CLINICAL TRIAL: NCT04268095
Title: Post Operative Dressing After Clean Elective Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Itay Ashkenazi (Other)
Responsible Party: Sponsor-Investigator, Itay Ashkenazi, Principal investigator, Tel Aviv Medical Center
Organization: Tel Aviv Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0548-18-TLV
Record Dates: First submitted 2020-02-05; First posted 2020-02-13 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Trigger Finger Disorder; Carpal Tunnel Syndrome; Ganglion
MeSH Terms: conditions — Trigger Finger Disorder; Carpal Tunnel Syndrome; Ganglion Cysts

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No dressing change (Experimental): Patients do not change dressing from procedure to first clinic followup after 14 days.
  Interventions: Other: Dressing protocol
- Ambulatory dressing change (Experimental): Patients change dressing by an ambulatory nurse (not associated with the study) 2 times a week from surgery to first clinic followup after 14 days
  Interventions: Other: Dressing protocol
- No dressing (Experimental): Patients take off dressing at post operative day 1 and clean it 3 times per day as instructed.
  Interventions: Other: Dressing protocol

INTERVENTIONS:
Other: Dressing protocol — Patients are assigned with different postoperative dressing protocols.

SUMMARY:
Very little has been published about the optimal post operative dressing protocol, and no practical conclusion has emerged from a meta-analysis published in 2013. Even fewer studies focused on that topic specifically in hand surgery. Nevertheless, the functional impairment due to a dressing in the hand is much greater than anywhere else, due to the constant use of hands in daily life activities. Yet, habits differs widely following surgeon's preference, from daily change with application of an antimicrobial unguent, to unchanged dressing until the first follow up consultation after 2 weeks, to complete removal of the dressing and basic soap and water cleaning at postoperative day (POD) 1. Those varying recommendations have functional and logistical implication for the patients, especially the elderlies, for whom autonomy is a fragile status that can be dramatically impaired by such protocols. The goal of this study is to define which post operative dressing protocol is optimal in terms of wound complications (disunion, infection)

ELIGIBILITY:
Inclusion Criteria:

* Elective hand surgery with clean wound (Type 1 in wound classification of american college of surgeon 11) - (Carpal tunnel, trigger finger, cyst removal or foreign body removal, tendon release).

Exclusion Criteria:

* Insertion of hardware
* Known skin condition disturbing normal healing,
* Immunodeficiency,
* Incapacity to understand or to observe the self cleaning protocol.
* Unexpected peroperative complication leading to a modification of the operative technique.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Instrumental activities of daily living questioner (IADL) | Baseline (Pre-op), 2 weeks, 6 weeks, 3 months
  Subjective function questioner. Scale 0-18. Higher score - better outcome.
Change in Vancouver Scar Scale | 2 weeks, 6 weeks, 3 months
  Evaluation of skin healing and scar formation. Scale 0-14. Higher score - inferior outcome.
Change in quick Disability of the Arm, Shoulder and Hand questioner (DASH) | Baseline, 2 weeks, 6 weeks, 3 months
  Subjective function questioner. Scale 0-100. Higher score - inferior outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv medical cemter, Tel Aviv, IL, Israel

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared at the discretion of the Chief Investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 30 days
Access Criteria: at the discretion of the Chief Investigator